CLINICAL TRIAL: NCT07048301
Title: Developing an Omaha System-Based Health Application on Improving Knowledge, Attitude, and Behaviors Regarding Infectious Disease Prevention in the Community
Brief Title: Omaha System-Based Health Application on Improving Knowledge, Attitude, and Behaviors Regarding Infectious Disease Prevention in the Community
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Atlas University (Other); Istanbul Medeniyet University (Other); Istanbul University - Cerrahpasa (Other); Hatay Devlet Hastanesi (Other); Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Gizemnur Torun, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-A4-01-39719
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Infectious Diseases; Attitude; Behavior; Knowledge
Keywords: Omaha System; Mobile health app
MeSH Terms: conditions — Communicable Diseases; Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUHOS app (Experimental): BUHOS app
  Interventions: Other: BUHOS app
- Control Group (Active Comparator): Control Group
  Interventions: Other: Control Group

INTERVENTIONS:
Other: BUHOS app — In this study, the BUHOS app initiative will be implemented among participants in the intervention group. BUHOS will be a two-weeks nursing intervention that includes monitoring KAB, employing Education, Guidance and Counseling (education videos), and Surveillance (reminder messages), and assessing the outcomes.
  Arms: BUHOS app
Other: Control Group — No intervention will be made to the patients in the control group, and the training videos prepared after the study is completed will be shared.
  Arms: Control Group

SUMMARY:
Background: Infectious diseases remain significant public health concerns due to several factors such as climate and environmental changes and natural disasters. Mobile health applications (mHealth apps) can be an appropriate way for fostering community participation, disseminating knowledge, and promoting behavior change toward infectious disease prevention. This study aims to describe a protocol for a pilot randomized controlled study to evaluate the impact of the Omaha System-Based mHealth app (BUHOS) on improving knowledge, attitude, and behaviors (KAB) regarding infectious disease prevention in an earthquake-affected region of Türkiye.

Methods: This study is a two-armed, parallel-group, randomized controlled trial design. A total of 112 eligible participants will be recruited from two separate container cities of an earthquake-affected region. These participants will be randomly allocated to either an intervention group or a control group. BUHOS will be designed based on the Omaha System, a widely recognized standardized taxonomy for the assessment, planning, and evaluation of healthcare services. BUHOS will be a two-week nursing intervention that includes monitoring KAB, employing Education, Guidance and Counseling (education videos), and Surveillance (reminder messages), and assessing the outcomes. Outcome variables will include the Problem Rating Scale for Outcomes, Community Communicable Diseases Knowledge Survey, Communicable Diseases Risk Awareness and Protection Scale and System Usability Scale. Outcome variables will be assessed on the 15th and 30th day after intervention.

Hypotheses:

H1: Among the Omaha System Problems, the Communicable/ Infectious Condition Problem Knowledge score will be higher on the 15th and 30th days compared to the control group.

H2: Infectious diseases risk awareness and prevention score will be higher on the 15th and 30th days compared to the control group.

H3: Communicable/ Infectious Condition Status Behaviour Parameter score will be higher on the 15th and 30th days compared to the control group H4: The knowledge and behaviour of the communicable/ infectious status and the awareness and prevention of the risk of infectious diseases of the experimental group will be higher than before the intervention on the 15th and 30th days.

ELIGIBILITY:
Inclusion criteria:

* being aged between 18 and 64 years,
* living in two container cities,
* having a knowledge score of 'very low (1)' and 'low (2)' on the Omaha System Problem Rating Scale for Outcome for Communicable/ Infectious Problem Knowledge Parameter,
* being literate,
* owning a smartphone.

Exclusion criteria:

* having impaired vision or hearing,
* having a mental illness,
* not owning a smartphone,
* being pregnant or postpartum,
* being participants in another scientific study,
* refusing to participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Omaha System- Problem Rating Scale for Outcomes Knowledge parameter | 15th and 30th day after intervention
Omaha System- Problem Rating Scale for Outcomes Behavior parameter | 15th and 30th day after intervention
Communicable Diseases Risk Awareness and Protection Scale (CDRAPS) | 15th and 30th day after intervention
Community Communicable Diseases Knowledge Survey | 15th and 30th day after intervention

SECONDARY OUTCOMES:
System Usability Scale (SUS) | 30th day after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin İlhan, Assoc. Prof., Principal Investigator — Istanbul Medeniyet University; Selda Seçginli, Study Director — Atlas University; Seda Doğru Bolat, Msc., Principal Investigator — Hatay State Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Secginli S, Altiner Yas M, Torun G, Ilhan N, Dogru Bolat S. Developing an Omaha System-based health application to improve knowledge, attitude, and behaviors regarding infectious disease prevention in the community: a study protocol for a randomized controlled trial. BMC Public Health. 2025 Nov 27;25(1):4170. doi: 10.1186/s12889-025-25587-8. PMID 41310526